CLINICAL TRIAL: NCT04239586
Title: Switching From Insulin to Sulfonylurea in Childhood and Adult Diabetes Due to Variants in the HNF1A, HNF4A, or HNF1B Genes
Brief Title: Switching From Insulin to Sulfonylurea in Diabetes Associated With Variants in MODY Genes
Acronym: SUtoChildT1D
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2388
Record Dates: First submitted 2020-01-02; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Maturity-Onset Diabetes of the Young, Type 3; Maturity Onset Diabetes of the Young, Type 1; Childhood Diabetes Mellitus; Insulin-dependent Diabetes Mellitus
Keywords: Maturity onset diabetes in the young; Childhood diabetes; Type 1 diabetes
MeSH Terms: conditions — Maturity-Onset Diabetes of the Young, Type 3; Maturity-Onset Diabetes of the Young, Type 1; Diabetes Mellitus, Type 1 | interventions — Sulfonylurea Compounds; Glyburide; Glipizide

STUDY DESIGN:
Intervention Model Description: Switching insulin-treated diabetes patients with possibly disease causing mutations in HNF1A, HNF4A, or HNF1B to treatment with sulfonylurea.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sulfonylurea treatment group (Experimental): Increasing doses of sulfonylurea class of drug to see whether insulin treatment can be reduced in dose or stopped.
  Interventions: Drug: Sulfonylurea

INTERVENTIONS:
Drug: Sulfonylurea — Starting treatment with sulfonylurea class of drug
  Other Names: Glibenclamide; Glipizide; Glimerepiride

SUMMARY:
The purpose of this study is to switch from insulin to oral sulfonylurea in patients with apparent type 1 diabetes or maturity onset diabetes in the young that are insulin treated. The molecular cause will be DNA variants in the HNF1A, HNF4A, or HNF1B genes that are of unknown significance (VUS, class 3) or known to be pathogenic (class 4 and 5).

DETAILED DESCRIPTION:
Maturity onset diabetes in the young (MODY) is characterised by monogenic diabetes due to beta-cell dysfunction, with typical onset of diabetes before age of 25 years. There are 14 known forms of MODY, ranging from rather common to extremely rare.

About 1% of patients in the Norwegian Childhood Diabetes registry may have disease causing MODY mutations, according to a study recently published by the investigator's group and others.

MODY associated mutations in the transcription factors HNF1A, HNF4A, and HNF1B leads to activation of the potassium channel causing depolarisation of the beta-cell membrane, which is crucial for excretion of insulin. By treating patients with HNF1A-MODY, HNF4A-MODY, and HNF1B-MODY with sulfonylurea class of drugs, these channels will close, causing depolarisation of the beta-cell membrane, and release of insulin. Hence, these patients can often stop insulin treatment when they are treated with sulfonylurea class drugs.

Due to high throughput sequencing, a number of rare variants in these genes have been discovered. In many cases, bioinformatic tools are not sufficient to correctly classify these variants. In the present study, we intend to identify rare variants in the HNF1A, HNF4A, and HNF1B genes in patients with insulin dependent diabetes identified through the Norwegian Childhood Diabetes registry or the Norwegian MODY Registry with possibly disease causing HNF1A, HNF4A, or HNF1B mutations with sulfonylurea to see if they can reduce or even stop insulin treatment, and regulate their diabetes with sulfonylurea only. All variants will be investigated by bioinformatics tools as well as functional assays (tests for DNA-binding, transcriptional activation, nuclear localisation, protein expression). Primary endpoints are efficacy of sulfonylurea treatment measured by insulin requirement or not and level of HbA1c. Secondary endpoints are tolerance of sulfonylurea and effect on insulin secretion by oral and intravenous glucose tolerance tests. Bioinformatics and functional characterisation will be compared with success to reach primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes and DNA sequence variant of unknown significance (VUS, class 3) or pathogenic (class 4, and 5) in the HNF1A, HNF4A, or HNF1B genes
* On insulin treatment
* Willing and able to provide informed consent (parents if younger than 16 years of age)

Exclusion Criteria:

* Known anaphylactic response to sulfonylurea
* Diabetes and DNA sequence variant in the HNF1A, HNF4A, or HNF1B genes that are known to be non-pathogenic (class 1-2)
* Not willing or able to provide informed consent (parents if younger than 16 years of age)

Ages: 2 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Effect of sulfonylurea treatment on insulin requirement measured in units insulin per kg per day | 5 years
  Effect of sulfonylurea treatment on insulin requirement measured in units insulin per kg bodyweight per day, recorded at intervals of 3-6 months after exposure to sulfonylurea compared to before initiation of sulfonylurea
Metabolic control of diabetes measured by HbA1c in mmol/mol | 5 years
  Metabolic control of diabetes measured by HbA1c in mmol/mol, recorded at intervals of 3-6 months after exposure to sulfonylurea compared to before initiation of sulfonylurea

SECONDARY OUTCOMES:
Level of sulfonylurea dose in mg per kg per day | 5 years
  Level of sulfonylurea dose in mg per kg body weight per day, recorded at intervals of 3-6 months after exposure to sulfonylurea compared to before initiation of sulfonylurea
Prevalence of side effects of sulfonylurea | 5 years
  Recording potential side effects of sulfonylurea, such as nausea, change in body weight, episodes of severe hypoglycemia, discolouration of teeth, diarrhoea, cardiovascular events, recorded at intervals of 3-6 months after exposure to sulfonylurea compared to before initiation of sulfonylurea
Effect on endogenous insulin secretion assessed by intravenous glucose tolerance tests | 5 years
  Maximum increment of serum insulin in nmol/L and serum c-peptide in pmol/L at intravenous glucose tolerance tests, recorded at intervals of 6-12 months after exposure to sulfonylurea compared to before initiation of sulfonylurea
Effect on secretion of incretin hormones, assessed by oral glucose tolerance tests | 5 years
  Maximum increment of serum insulin in nmol/L, serum c-peptide in pmol/L and incretins (GIP in pmol/L and GLP-1 in pmol/L) at oral glucose tolerance tests and in comparison with intravenous gluclose tolerance tests, recorded at intervals of 6-12 months after exposure to sulfonylurea compared to before initiation of sulfonylurea

CONTACTS AND LOCATIONS:
Overall Officials: Pål R. Njølstad, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Department of Pediatrics and Adolescents, Haukeland University Hospital, and Department of Clinical Science, Faculty of Medicine, University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results in the planned publications. The IPD will be summary data, and with no personal identifiers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the planned publications are finally accepted for publication.
Access Criteria: IPD will be shared after written request and consideration to the corresponding author of the respective publication. Data will be shared with researchers in the same or similar field only. IPD will include summary data without personal identity and Describe by what access criteria IPD and any additional supporting information will be shared, including with whom, for what types of analyses, and by what mechanism. The corresponding and first authors will review requests and criteria for reviewing requests may also be provided.

REFERENCES:
- [Background] Gloyn AL, Pearson ER, Antcliff JF, Proks P, Bruining GJ, Slingerland AS, Howard N, Srinivasan S, Silva JM, Molnes J, Edghill EL, Frayling TM, Temple IK, Mackay D, Shield JP, Sumnik Z, van Rhijn A, Wales JK, Clark P, Gorman S, Aisenberg J, Ellard S, Njolstad PR, Ashcroft FM, Hattersley AT. Activating mutations in the gene encoding the ATP-sensitive potassium-channel subunit Kir6.2 and permanent neonatal diabetes. N Engl J Med. 2004 Apr 29;350(18):1838-49. doi: 10.1056/NEJMoa032922. PMID 15115830
- [Background] Sagen JV, Raeder H, Hathout E, Shehadeh N, Gudmundsson K, Baevre H, Abuelo D, Phornphutkul C, Molnes J, Bell GI, Gloyn AL, Hattersley AT, Molven A, Sovik O, Njolstad PR. Permanent neonatal diabetes due to mutations in KCNJ11 encoding Kir6.2: patient characteristics and initial response to sulfonylurea therapy. Diabetes. 2004 Oct;53(10):2713-8. doi: 10.2337/diabetes.53.10.2713. PMID 15448106
- [Background] Pearson ER, Flechtner I, Njolstad PR, Malecki MT, Flanagan SE, Larkin B, Ashcroft FM, Klimes I, Codner E, Iotova V, Slingerland AS, Shield J, Robert JJ, Holst JJ, Clark PM, Ellard S, Sovik O, Polak M, Hattersley AT; Neonatal Diabetes International Collaborative Group. Switching from insulin to oral sulfonylureas in patients with diabetes due to Kir6.2 mutations. N Engl J Med. 2006 Aug 3;355(5):467-77. doi: 10.1056/NEJMoa061759. PMID 16885550
- [Background] Rafiq M, Flanagan SE, Patch AM, Shields BM, Ellard S, Hattersley AT; Neonatal Diabetes International Collaborative Group. Effective treatment with oral sulfonylureas in patients with diabetes due to sulfonylurea receptor 1 (SUR1) mutations. Diabetes Care. 2008 Feb;31(2):204-9. doi: 10.2337/dc07-1785. Epub 2007 Nov 19. PMID 18025408
- [Background] Stoffers DA, Zinkin NT, Stanojevic V, Clarke WL, Habener JF. Pancreatic agenesis attributable to a single nucleotide deletion in the human IPF1 gene coding sequence. Nat Genet. 1997 Jan;15(1):106-10. doi: 10.1038/ng0197-106. PMID 8988180
- [Background] Njolstad PR, Sovik O, Cuesta-Munoz A, Bjorkhaug L, Massa O, Barbetti F, Undlien DE, Shiota C, Magnuson MA, Molven A, Matschinsky FM, Bell GI. Neonatal diabetes mellitus due to complete glucokinase deficiency. N Engl J Med. 2001 May 24;344(21):1588-92. doi: 10.1056/NEJM200105243442104. No abstract available. PMID 11372010
- [Background] Babenko AP, Polak M, Cave H, Busiah K, Czernichow P, Scharfmann R, Bryan J, Aguilar-Bryan L, Vaxillaire M, Froguel P. Activating mutations in the ABCC8 gene in neonatal diabetes mellitus. N Engl J Med. 2006 Aug 3;355(5):456-66. doi: 10.1056/NEJMoa055068. PMID 16885549
- [Background] Johansson BB, Irgens HU, Molnes J, Sztromwasser P, Aukrust I, Juliusson PB, Sovik O, Levy S, Skrivarhaug T, Joner G, Molven A, Johansson S, Njolstad PR. Targeted next-generation sequencing reveals MODY in up to 6.5% of antibody-negative diabetes cases listed in the Norwegian Childhood Diabetes Registry. Diabetologia. 2017 Apr;60(4):625-635. doi: 10.1007/s00125-016-4167-1. Epub 2016 Dec 2. PMID 27913849
- [Background] Irgens HU, Molnes J, Johansson BB, Ringdal M, Skrivarhaug T, Undlien DE, Sovik O, Joner G, Molven A, Njolstad PR. Prevalence of monogenic diabetes in the population-based Norwegian Childhood Diabetes Registry. Diabetologia. 2013 Jul;56(7):1512-9. doi: 10.1007/s00125-013-2916-y. Epub 2013 Apr 27. PMID 23624530
- [Background] Najmi LA, Aukrust I, Flannick J, Molnes J, Burtt N, Molven A, Groop L, Altshuler D, Johansson S, Bjorkhaug L, Njolstad PR. Functional Investigations of HNF1A Identify Rare Variants as Risk Factors for Type 2 Diabetes in the General Population. Diabetes. 2017 Feb;66(2):335-346. doi: 10.2337/db16-0460. Epub 2016 Nov 29. PMID 27899486
- [Background] Hattersley AT, Greeley SAW, Polak M, Rubio-Cabezas O, Njolstad PR, Mlynarski W, Castano L, Carlsson A, Raile K, Chi DV, Ellard S, Craig ME. ISPAD Clinical Practice Consensus Guidelines 2018: The diagnosis and management of monogenic diabetes in children and adolescents. Pediatr Diabetes. 2018 Oct;19 Suppl 27:47-63. doi: 10.1111/pedi.12772. No abstract available. PMID 30225972
- [Background] Bowman P, Sulen A, Barbetti F, Beltrand J, Svalastoga P, Codner E, Tessmann EH, Juliusson PB, Skrivarhaug T, Pearson ER, Flanagan SE, Babiker T, Thomas NJ, Shepherd MH, Ellard S, Klimes I, Szopa M, Polak M, Iafusco D, Hattersley AT, Njolstad PR; Neonatal Diabetes International Collaborative Group. Effectiveness and safety of long-term treatment with sulfonylureas in patients with neonatal diabetes due to KCNJ11 mutations: an international cohort study. Lancet Diabetes Endocrinol. 2018 Aug;6(8):637-646. doi: 10.1016/S2213-8587(18)30106-2. Epub 2018 Jun 4. PMID 29880308
- [Background] Sagen JV, Bjorkhaug L, Haukanes BI, Grevle L, Molnes J, Nedrebo BG, Sovik O, Njolstad PR, Johansson S, Molven A. The HNF1A mutant Ala180Val: Clinical challenges in determining causality of a rare HNF1A variant in familial diabetes. Diabetes Res Clin Pract. 2017 Nov;133:142-149. doi: 10.1016/j.diabres.2017.08.001. Epub 2017 Sep 1. PMID 28934671
- [Background] Flannick J, Johansson S, Njolstad PR. Common and rare forms of diabetes mellitus: towards a continuum of diabetes subtypes. Nat Rev Endocrinol. 2016 Jul;12(7):394-406. doi: 10.1038/nrendo.2016.50. Epub 2016 Apr 15. PMID 27080136
- [Background] Balamurugan K, Bjorkhaug L, Mahajan S, Kanthimathi S, Njolstad PR, Srinivasan N, Mohan V, Radha V. Structure-function studies of HNF1A (MODY3) gene mutations in South Indian patients with monogenic diabetes. Clin Genet. 2016 Dec;90(6):486-495. doi: 10.1111/cge.12757. Epub 2016 Mar 4. PMID 26853433
- [Background] Flannick J, Beer NL, Bick AG, Agarwala V, Molnes J, Gupta N, Burtt NP, Florez JC, Meigs JB, Taylor H, Lyssenko V, Irgens H, Fox E, Burslem F, Johansson S, Brosnan MJ, Trimmer JK, Newton-Cheh C, Tuomi T, Molven A, Wilson JG, O'Donnell CJ, Kathiresan S, Hirschhorn JN, Njolstad PR, Rolph T, Seidman JG, Gabriel S, Cox DR, Seidman CE, Groop L, Altshuler D. Assessing the phenotypic effects in the general population of rare variants in genes for a dominant Mendelian form of diabetes. Nat Genet. 2013 Nov;45(11):1380-5. doi: 10.1038/ng.2794. Epub 2013 Oct 6. PMID 24097065
- [Derived] Svalastoga P, Kaci A, Molnes J, Solheim MH, Johansson BB, Krogvold L, Skrivarhaug T, Valen E, Johansson S, Molven A, Sagen JV, Softeland E, Bjorkhaug L, Tjora E, Aukrust I, Njolstad PR. Characterisation of HNF1A variants in paediatric diabetes in Norway using functional and clinical investigations to unmask phenotype and monogenic diabetes. Diabetologia. 2023 Dec;66(12):2226-2237. doi: 10.1007/s00125-023-06012-4. Epub 2023 Oct 5. PMID 37798422